CLINICAL TRIAL: NCT03006016
Title: Impact of Preoperative 4-week Supplementation With Omega-3 Polyunsaturated Fatty Acids on Liver Volume and Steatosis to Facilitate Bariatric Surgery in Morbdly Obese Patients : the " Omegaobese Study ".
Brief Title: Preoperative Omega-3 Polyunsaturated Fatty Acids in Morbidly Obese to Reduce Liver Volume and Steatosis
Acronym: Omegobese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-API-03
Record Dates: First submitted 2016-12-08; First posted 2016-12-30 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2021-09

CONDITIONS: Morbid Obesity D009765
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 (Experimental): The patient will take Omega 3 before intervention 4-week course of 1.500 Mg/ day without caloric restriction
  Interventions: Drug: Omega-3 Fatty Acid
- Placebo (Placebo Comparator): The patient will take placebo before intervention 4-week course of 1.500 Mg/ day without caloric restriction
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omega-3 Fatty Acid — The enrollment in the study is proposed by an investigator (surgeon) in each centre at the time of a preoperative visit (V0). Randomization takes place the week before the visit with the investigating surgeon in charge of the patient (V1) when the bariatric procedure is scheduled: omega-3 group (1650 mg of omega-3 / day for 4 weeks without caloric restriction) or placebo group.
  Arms: Omega 3
Other: Placebo — The enrollment in the study is proposed by an investigator (surgeon) in each centre at the time of a preoperative visit (V0). Randomization takes place the week before the visit with the investigating surgeon in charge of the patient (V1) when the bariatric procedure is scheduled: omega-3 group (1650 mg of omega-3 / day for 4 weeks without caloric restriction) or placebo group.
  Arms: Placebo

SUMMARY:
Hepatomegaly is common in the morbidly obese patients and it may hamper the access to the hiatal region during bariatric surgery. The doctors made a preliminary prospective study that showed that a preoperative 4-week course of 1.500 Mg/ day without caloric restriction resulted in a 20 % reduction in the volume of the left liver lobe (segment 2 and 3) on ultrasounds.

The aim of this study is to determine whether a 4-week preoperative course with omega-3 without caloric restriction (1650 mg of omega-3 / day for 4 weeks) may reduce liver volume and its fat content, rendering thus surgery easier.

The primary end point is the reduction of the volume of the left liver lobe as measured by magnetic resonance imaging.

Secondary end points are: the reduction of the whole liver volume, liver steatosis, liver injuries during surgery, and duration of surgery, the evolution of liver tests as well as the correlation between preoperative MRI data and intraoperative liver biopsy for the quantification of liver steatosis.

Study design: This is an interventional, prospective, multicentric, randomized, double blinded clinical trial. Morbidly obese patients with metabolic syndrome candidate to bariatric surgery fulfilling criteria for bariatric surgery as established by the Haute Autorité de Santé are elegible for the study. Number of subjects to be enrolled: 44 patients in 12 months.

Study time schedule: At the time of the enrollment visit two visits are scheduled, the first before the beginning of the study and the last at the end. Surgery is scheduled no more than 7 days after the end of the treatment. At time of these two visits a clinical examination is performed avec calculation of the BMI, blood tests (ASAT, ALAT; GGT, total, HDL and LDL cholesterol, triglycerides, glycemia, C-peptide, HbA1c, insulin, HOMA-IR, C reactive protein) and a MRI to evaluate the volume and the fat content of the liver. At time of surgery duration of surgery and any eventual liver injury are recorded and a liver biopsy is performed.

The hypothesis is that, as shown by the preliminary study, the omega-3, will result in a reduction in the volume of the left liver lobe of 20 %.

Conclusion: If a 4-week preoperative course of omega-3 without caloric restriction results in a significant reduction of liver volume and steatosis before bariatric surgery, it may be recommended as a systematic preoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* Karnofsky Index de > 70
* BMI > 35 kg/m2 associated with metabolic syndrome define by three or more of the following: waistline that measures at least 80 centimeters for european women and 94 centimeters for european men; High triglyceride level less than 1.5 g/l or specific medications; Reduced high-density lipoprotein (HDL) cholesterol less than 1.04 mmol/L in men or less than 1.3 mmol/L in women; Increased blood pressure 130/85 millimeters of mercury (mm Hg) or higher or specific medications; Elevated fasting blood sugar 100 mg/dL (5.6 mmol/L) or higher or specific médications.
* Failure of previous medical treatment of morbid obesity well conducted by a multidisciplinary team for at least 6 months.
* Multidisciplinary team agreement for bariatric surgery
* Patients affiliated to the French Health Care System (Sécurité Sociale)
* Patients having signed the informed consent

Exclusion Criteria:

* Contraindications to MRI (pace-maker, metallic foreign bodies, claustrophobia)
* Psychiatric contraindications to bariatric surgery
* Anesthesiology contraindications to surgery
* Progressive malignancies
* Chronic alcoholism (>30 gr/day)
* Uncontrolled sepsis
* History of liver disease
* Renal failure (Cockroft <30ml/min)
* Long term treatment with steroids
* Regular assumption of alimentary complements enriched with proteins and/or amino acids)
* Pregnancy (pregnancy test will be done before surgery in fertile women)
* History of bariatric surgery of supramesocolic surgery rendering the access to the hiatal region difficult.
* Forseeable difficulies in completing follow-up
* Patients under judicial protection
* Patients unable to understand or put in practice medical prescription as omega-3 oral supplementation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
The volume of the left liver lobe | 4 weeks
  Reduction of the volume of the left liver lobe as measured by magnetic resonance imaging between the beginning of the study and its end (4 weeks)

SECONDARY OUTCOMES:
The whole liver volume | 4 weeks
  Reduction of the whole liver volume (as measured on MRI)
The liver injuries | 4 weeks
  liver injuries during surgery (surgeon report)

OTHER OUTCOMES:
the liver steatosis | 4 weeks
  Reduction of the whole liver steatosis (as measured on MRI)

CONTACTS AND LOCATIONS:
Overall Officials: IANNELLI Antonio, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CHU de Nice - Chirurgie Digestive- Hôpital Archet, Nice, Alpes-maritimes
  - CHU de Montpellier - Chirurgie digestive, Montpellier, Languedoc - Roussillon

IPD SHARING:
Plan to Share IPD: No